CLINICAL TRIAL: NCT00050531
Title: Randomized Trial of Therapy of Early Phase Chronic Myelogenous Leukemia With High-Dose Imatinib Mesylate (Gleevec) Alone or in Combination With Peg-Alpha Interferon (PEG-Intron) and Sargramostim (GM-CSF)
Brief Title: High-Dose Gleevec Alone or in Combination With Peg-Intron and GM-CSF in Early Phase Chronic Myelogenous Leukemia (CML)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ID02-534; NCI-2012-01295 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2002-12-12; First posted 2003-02-07 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2015-08

CONDITIONS: Leukemia, Myeloid, Chronic
Keywords: Chronic Myelogenous Leukemia; CML; Early Chronic Phase Chronic Myelogenous Leukemia; Imatinib Mesylate; Gleevec; Peg-Alpha Interferon; Peg-Intron; Sargramostim; GM-CSF
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Myeloid, Chronic-Phase | interventions — Imatinib Mesylate; peginterferon alfa-2b; Interferon alpha-2; sargramostim; Granulocyte-Macrophage Colony-Stimulating Factor; Colony-Stimulating Factors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Gleevec (Experimental): Gleevec 400 mg orally twice daily.
  Interventions: Drug: Gleevec; Drug: Peg-alpha interferon (Peg-Intron)
- Gleevec + Peg-Intron + GM-CSF (Experimental): Gleevec 400 mg orally twice daily. Peg-Intron 0.5 mcg/kg each week subcutaneously. GM-CSF 125 mcg/m^2 three times per week subcutaneously.
  Interventions: Drug: Gleevec; Drug: Peg-alpha interferon (Peg-Intron); Drug: Sargramostim (GM-CSF)

INTERVENTIONS:
Drug: Gleevec — 400 mg orally twice daily.
  Other Names: Imatinib Mesylate; STI-571
Drug: Peg-alpha interferon (Peg-Intron) — PEG-IFN 0.5 mcg/kg each week subcutaneously.
  Other Names: PEG Interferon; Interferon Alfa-2b (PEG conjugate)
Drug: Sargramostim (GM-CSF) — 125 mcg/m^2 three times per week subcutaneously.
  Other Names: LeukineTM; Granulocyte-Macrophage Colony Stimulating Factor
  Arms: Gleevec + Peg-Intron + GM-CSF

SUMMARY:
The goal of this clinical research study is to learn if giving PEG-Alpha Interferon (PEG-Intron) and Sargramostim (GM-CSF) to patients receiving treatment with high dose Gleevec (imatinib mesylate) is more effective in treating CML in chronic phase than therapy with imatinib mesylate alone.

DETAILED DESCRIPTION:
Imatinib mesylate is a drug that blocks a protein that is responsible for the development of CML. PEG-Intron is a natural substance made by the cells of the immune system and helps to control CML. GM-CSF is a hormone that helps to stimulate the production of white blood cells.

During the study you will take 400 mg of imatinib mesylate by mouth 2 times a day (800 mg a day total). Imatinib mesylate should be taken each morning and evening with a large glass of water. You may be given a "pill diary" to write down when (day and time) you take the drug. You may also write in the diary any side effects you may experience. You may bring the diary, any unused tablets, and empty bottles of imatinib mesylate with you to every visit to the study doctor. Any unused supplies must be returned at the end of the study.

After completing 6 months of imatinib mesylate therapy, you will be randomly assigned (as in the toss of a coin) to one of two groups. Patients in the first group will be given PEG-Intron and GM-CSF in addition to imatinib mesylate therapy. Patients in the other group will continue taking only imatinib mesylate.

If you are assigned to the group that will receive PEG-Intron and GM-CSF, you will continue taking imatinib mesylate. In addition, PEG-Intron will be given as an injection under the skin once a week. Sargramostim will be given as an injection under the skin 3 times a week. You and/or your family members can be taught to give these injections.

Every 1-2 weeks during the first 4 weeks of the study, you will have around 2 teaspoons of blood drawn for routine blood tests and to measure the amount of imatinib in your blood. The blood tests will then be repeated every 6 to 8 weeks (or more often if your doctor feels it is necessary) for as long as you are on the study. A bone marrow sample will also be taken every 3 months for the first year and then every 4 to 6 months for as long as you are on the study to check on the status of the disease .

You will be asked to visit the doctor for a physical exam and to have vital signs measured. These visits will be scheduled at least every 3 months while you are on the study. The visits may be scheduled more often depending on the status of the disease.

Update: February 2012:

Blood test are recommended 2 times per year. Your doctor will discuss with you how often you should have blood tests. Bone marrow will be done if your doctor thinks it is needed to check the disease. You must return to M.D. Anderson at least once every year. You may not need a bone marrow test every visit, but you will have blood drawn to measure the amount of disease you have.

Treatment in both groups may be continued for up to 7-10 years, or as long as the doctor feels is necessary to control the leukemia.

If the disease gets worse or you experience any intolerable side effects, you will be taken off the study and your doctor will discuss other treatment options with you.

This is an investigational study. All of the drugs used in this study are FDA approved and commercially available. However, their use in this study is investigational. A total of 98 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with Ph-positive CML in early chronic phase CML who have received no or minimal prior therapy, (<1 month of prior IFN-alpha (with or without ara-C) and/or Gleevec).
2. Eastern Cooperative Oncology Group (ECOG) performance of 0-2.
3. Adequate end organ function, defined as the following: total bilirubin < 1.5 x upper limit of normal (ULN), serum glutamate pyruvate transaminase (SGPT) < 2.5 x ULN, creatinine < 1.5 x ULN
4. Signed informed consent.

Exclusion Criteria:

1. New York Heart Association (NYHA) cardiac class 3-4 heart disease.
2. Psychiatric disability (psychosis)
3. Pregnant or lactating females
4. Late chronic phase, accelerated or blastic phase

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2003-04; Primary Completion 2007-04 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Duration of Pathological Complete Response Negativity or Cytogenetic Response | Molecular response at 12 Months and Polymerase Chain Reaction (PCR) testing once a year (+/- 3 months)
  Duration measured in time from first response to disease progression; Cytogenetic (or FISH), and PCR quantification every 3-4 months as indicated in year one then FISH every 1-3 years and PCR every year
Number of Participants with Complete Hematologic Remission (CHR) Classification of Complete Cytogenetic Response | Molecular response at 12 Months
  Complete Hematologic Remission (CHR) - normalization >4 weeks of bone marrow (less than 5% blasts) & peripheral blood with white blood count (WBC)<10x10^9/L & no peripheral blasts, promyelocytes or myelocytes, disappearance of all signs & symptoms of disease. Partial Hematologic Response (PHR) = CHR except persistence of immature cells (myelocytes, metamyelocytes), or splenomegaly <50% of pretreatment, or thrombocytosis >450x10^9/L but <50% of pretreatment. Complete hematologic remission further classified according to suppression of Philadelphia chromosome (Ph) by cytogenetics or fluorescence in situ hybridization (FISH): a) No cytogenetic response - Ph positive 100% of pretreatment value; b) Minor cytogenetic response - Ph positive 35-90% of pretreatment value; c) Partial cytogenetic response - Ph positive 1-34% of pretreatment value; d) Complete cytogenetic response - Ph positive 0%.

CONTACTS AND LOCATIONS:
Overall Officials: Jorge E Cortes, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Jain P, Kantarjian H, Boddu PC, Nogueras-Gonzalez GM, Verstovsek S, Garcia-Manero G, Borthakur G, Sasaki K, Kadia TM, Sam P, Ahaneku H, O'Brien S, Estrov Z, Ravandi F, Jabbour E, Cortes JE. Analysis of cardiovascular and arteriothrombotic adverse events in chronic-phase CML patients after frontline TKIs. Blood Adv. 2019 Mar 26;3(6):851-861. doi: 10.1182/bloodadvances.2018025874. PMID 30885996
- [Derived] Issa GC, Kantarjian HM, Gonzalez GN, Borthakur G, Tang G, Wierda W, Sasaki K, Short NJ, Ravandi F, Kadia T, Patel K, Luthra R, Ferrajoli A, Garcia-Manero G, Rios MB, Dellasala S, Jabbour E, Cortes JE. Clonal chromosomal abnormalities appearing in Philadelphia chromosome-negative metaphases during CML treatment. Blood. 2017 Nov 9;130(19):2084-2091. doi: 10.1182/blood-2017-07-792143. Epub 2017 Aug 23. PMID 28835440
- [Derived] Jain P, Kantarjian H, Nazha A, O'Brien S, Jabbour E, Romo CG, Pierce S, Cardenas-Turanzas M, Verstovsek S, Borthakur G, Ravandi F, Quintas-Cardama A, Cortes J. Early responses predict better outcomes in patients with newly diagnosed chronic myeloid leukemia: results with four tyrosine kinase inhibitor modalities. Blood. 2013 Jun 13;121(24):4867-74. doi: 10.1182/blood-2013-03-490128. Epub 2013 Apr 25. PMID 23620574
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org